CLINICAL TRIAL: NCT05739032
Title: Exercise Training Six-Months After Discharge in Post-COVID-19 Syndrome: Randomized Controlled Trial
Brief Title: Exercise Training Six-Months After Discharge in Post-COVID-19 Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ukbe Sirayder (Other)
Responsible Party: Sponsor-Investigator, Ukbe Sirayder, Principal Investigator, Nuh Naci Yazgan University
Organization: Nuh Naci Yazgan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNYUSİRAYDER1
Record Dates: First submitted 2023-02-21; First posted 2023-02-22 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: COVID-19 Pneumonia
Keywords: post-COVID-19; Lung function; Fatigue; Aerobic exercise; Strength training
MeSH Terms: conditions — Fatigue | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Exercise group received aerobic exercise (30-min walking) and upper and lower extremity strength training for 12 weeks for 3 days/week.
  Interventions: Other: Aerobic exercise and strength training
- Control group (No Intervention): Control group continued only routine follow-up.

INTERVENTIONS:
Other: Aerobic exercise and strength training — Aerobic Exercise Training: The individuals in the study group were given aerobic exercise training at 70-80% of the 6MWT average speed. Patients performed exercise three days per week (twice under the supervision of a physiotherapist and once at home) for 30 minutes a day.
  Strength Training: Lower and upper extremity strengthening training was performed three days a week, 3x10-12 repetitions per day, with the help of a resistance band suitable for muscle strength. Hip flexion, hip abduction, knee flexion, and knee extension exercises for the lower extremity, and shoulder flexion, shoulder extension, shoulder abduction, shoulder elevation, external rotation, horizontal shoulder abduction, and scapular adduction exercises for the upper extremity were performed.
  Arms: Exercise group

SUMMARY:
The goal of this study investigate the effects of 12-week exercise training on pulmonary function, symptoms, functional capacity, and quality of life (QoL) in patients with severe COVID 6 months after intensive care discharge. The main question it aims to answer are:

1-Does exercise training given in post-COVID-19 syndrome have an effect on pulmonary function, symptoms, functional capacity, muscle strength and quality of life?

25 severe post-COVID patients (35 M) were in exercise group (EG) (age=52.9±11 years, 18M), and 25 (age=53.6±11.9 years, 17M) were in the control group (CG). EG received aerobic exercise (30-min walking) and upper and lower extremity strength training for 12 weeks for 3 days/week. CG continued only routine follow-up.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 pneumonia patients were followed up for at least 24 h in the ICU. Those post-COVID six months who could cooperate with the tests and volunteered to participate were included.

Exclusion Criteria:

* Individuals with pulmonary, orthopedic, neurological, vestibular, and psychological problems diagnosed before COVID-19 infection; myocarditis developed after COVID-19 infection; and those pregnant and those having any other acute diseases (such as infection and trauma) that would prevent performing the tests and/or interfering with the test results were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Test Distance | six minute

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
send via mail
Supporting Information: Study Protocol, SAP, CSR
Time Frame: two years